CLINICAL TRIAL: NCT06263283
Title: Impact of an Educational Physiotherapy-Yoga Intervention on Perceived Stress in Women Treated With Brachytherapy for Cervical Cancer: a Randomized Controlled Trial
Brief Title: Impact of an Educational Physiotherapy-Yoga Intervention on Perceived Stress in Women Treated With Brachytherapy for Cervical Cancer
Acronym: KYOCOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2023-04 KYO
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cervical Cancer; Brachytherapy
Keywords: cervical cancer; uterovaginal brachytherapy; stress; Prolonged immobilization; yoga
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Control Group: Standard care according to the modalities of each center (concomitant treatment prescription, psychological support, physiotherapy or dietetic are supports that can be proposed if needed) Experimental Group: Standard support with Daily realization of a session of Kine-Yoga supervised by a physiotherapist at J2, J3 and J4 of uterovaginal brachytherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard care according to the modalities of each center (concomitant treatment prescription, psychological support, physiotherapy or dietetic are supports that can be proposed if needed)
- Experimental Group (Experimental): Standard support with Daily realization of a session of Kine-Yoga supervised by a physiotherapist at J2, J3 and J4 of uterovaginal brachytherapy.
  Possibility for the patient to practice this session in autonomy (using PEP tools given to the Shared Educational Check-up) according to her wish during the duration of the treatment and up to 15 days post treatment.
  Interventions: Other: session of Kine-Yoga

INTERVENTIONS:
Other: session of Kine-Yoga — Daily performance of a Kine-Yoga-PEP intervention supervised by a physiotherapist of the department trained in the Kine-Yoga-PEP intervention at J2, J3 and J4 of uterovaginal brachytherapy.
  Possibility for the patient to practice this session in autonomy (using PEP tools given to the Shared Educational Check-up) according to her wish during the duration of the treatment and up to 15 days post treatment
  Arms: Experimental Group

SUMMARY:
Every year in France, nearly 3,000 women develop a cervical cancer. The average age of women diagnosed is 51. Uterovaginal brachytherapy is one of the reference treatments.

To allow this treatment, an applicator is first placed under general anaesthesia in the vaginal zone. Then, the pulsed Dose Rate (PDR) or high dose rate (HDR) uterovaginal brachytherapy requires 2-5 days hospitalization in an isolated room. Uterovaginal brachytherapy requires strict bed rest without movements allowed for the pelvic area until the applicator is removed.

Prolonged immobilization, the context of the illness and the intimacy of the area to be treated are all recognized sources of anxiety. According to a study, 40% of patients have post-traumatic stress at 3 months of treatment. A Danish team highlights the significant decrease in physical capacity during and after treatment.

Thus, as a recent literature review concludes, there is a real need to develop Non-Pharmacological-Interventions (NPI) to limit the aftereffects. It also seems important to provide support for self-management of symptoms.

Among NPI of interest, Yoga is a mind-body practice that can decrease perceived stress. A systematic review confirms that yoga can reduce stress during cancer treatment. This underlines the importance of proposing this practice for patients treated for all types of cancers and further evaluations on the effects of respiratory and meditation exercises. Another team showed the feasibility of respiratory exercise intervention in patients undergoing chemotherapy while also talking about mental health benefits. Finally, a reduction in perceived stress was achieved in women treated with radiotherapy for breast cancer through yoga intervention. A lot of work has been done with promising results without the result of a consensus applicable to all care situations.

Moreover, educational requirements are high in women treated to gynecological cancer.

Meeting these needs helps to improve quality of life, pain management and drug use.

Integrating Patient Educational Project (PEP) therefore seems relevant as an additional tool in patient empowerment. In addition, the fact that a combined Physiotherapy-Yoga-PEP intervention is feasible in women treated for breast cancer allows us to offer adjusted version in patients with brachytherapy.

The literature review thus invites us to propose the educational intervention Kine-Yoga-PEP in the very particular context of brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Woman 18 ≥ years old, no age limit
* Patient treated for cervical cancer (histologically proven) by uterovaginal brachytherapy
* Patient with stress level ≥ 3 on VAS from 0 to 10
* Patient´s signed written informed consent
* Affiliation to a French Social Security System

Exclusion Criteria:

* Physical alteration not allowing the practice of Yoga,
* Patient does not understand and does not speak French
* Patient whose regular follow-up is initially impossible for psychological, family, social or geographical reasons,
* Patient under guardianship or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Kine-Yoga-PEP intervention to standard care during the uterovaginal brachytherapy on perceived stress at 15 days of treatment initiation in patients treated for cervical cancer. | Time from the randomization to 15 days after uterovaginal brachytherapy
  The Perceived Stress Score will be assessed by the 10-item Perceived Stress Scale (PSS) self-assessment 15 days after the start of the uterovaginal brachytherapy.

SECONDARY OUTCOMES:
assessment in the experimental group: safety and patient compliance at the Kine-Yoga-PEP intervention | Time from the randomization to 15 days after uterovaginal brachytherapy
  The safety will be evaluated by Number of treatment interruptions due to applicator displacement and/or source friction following Kine-Yoga-PEP intervention. Patient compliance will be evaluated by the number of sessions performed (supervised and independent) collected on the logbooks filled out by the patients
Evaluation of the immediate effect of the Kine-Yoga-PEP intervention in the experimental group on perceived stress, pain (overall and due to immobility) and the evolution of these parameters during brachytherapy. | During the uterovaginal brachytherapy.
  Scores obtained at the Visual Analog Scales (VAS) of stress and EVA of pain (global and immobility-related), before and after Kine-Yoga-PEP intervention and during uterovaginal brachytherapy.
Evaluation of the evolution of fatigue during uterovaginal brachytherapy | During the uterovaginal brachytherapy.
  Fatigue score obtained on Visual Analogue Scale (VAS) during uterovaginal brachytherapy
assessment of the psychological distress at inclusion and 15 days after the uterovaginal brachytherapy | Time from the baseline to 15 days after uterovaginal brachytherapy
  Anxiety-Depressive Distress Score measured by the Hospital Anxiety and Depression Scale (HADS) Questionnaire for uterovaginal Brachytherapy at inclusion and 15 days after the uterovaginal brachytherapy
Description of the use of anxiolytics by group (experimental vs control) | Time from the baseline to 15 days after uterovaginal brachytherapy
  The use of anxiolytic treatments will be described in the logbooks filled out by the patients
Description of the experiences of patients treated for cervical cancer during uterovaginal brachytherapy receiving a Kine-Yoga-PEP intervention (approximately 20 patients in the experimental group | Between 7 or 12 days after the uterovaginal brachytherapy
  The diversity of verbatim and semantic themes collected by a 40 - 60 minute semi-directional interview (qualitative analysis) in the week following the removal of the applicator from patients until data saturation (approximately 20 patients in the experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Aurore MOUSSION, Study Director — INSTITUT REGIONAL DU CANCER DE MONTPELLIER Cancer de Montpellier; Kerstin FARAVEL, Principal Investigator — INSTITUT REGIONAL DU CANCER DE MONTPELLIER Cancer de Montpellier
Locations (3):
- France (3):
  - ICM, Montpellier
  - Centre Eugène Marquis, Rennes
  - Oncopole Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after encoding with an inclusion number, 1st letter of the name and surname may be shared.
  The data of the participants will be available upon request and with the completion of a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan (PAS) and the analytical code may also be subject to data sharing as part of a transfer contract (RGPD)

REFERENCES:
- [Background] Booth K, Beaver K, Kitchener H, O'Neill J, Farrell C. Women's experiences of information, psychological distress and worry after treatment for gynaecological cancer. Patient Educ Couns. 2005 Feb;56(2):225-32. doi: 10.1016/j.pec.2004.02.016. PMID 15653253
- [Background] Kirchheiner K, Czajka-Pepl A, Ponocny-Seliger E, Scharbert G, Wetzel L, Nout RA, Sturdza A, Dimopoulos JC, Dorr W, Potter R. Posttraumatic stress disorder after high-dose-rate brachytherapy for cervical cancer with 2 fractions in 1 application under spinal/epidural anesthesia: incidence and risk factors. Int J Radiat Oncol Biol Phys. 2014 Jun 1;89(2):260-7. doi: 10.1016/j.ijrobp.2014.02.018. Epub 2014 Apr 7. PMID 24721589
- [Background] Holt KA, Mogensen O, Jensen PT, Hansen DG. Goal setting in cancer rehabilitation and relation to quality of life among women with gynaecological cancer. Acta Oncol. 2015 Nov;54(10):1814-23. doi: 10.3109/0284186X.2015.1037009. Epub 2015 May 6. PMID 25943136
- [Background] Humphrey P, Bennett C, Cramp F. The experiences of women receiving brachytherapy for cervical cancer: A systematic literature review. Radiography (Lond). 2018 Nov;24(4):396-403. doi: 10.1016/j.radi.2018.06.002. Epub 2018 Jul 18. PMID 30292512
- [Background] Christiansen MG, Piil K, Jarden M. The Symptom Experience and Self-management Strategies of Women Undergoing Cervical Cancer Treatment: A Qualitative Study. Cancer Nurs. 2022 Jan-Feb 01;45(1):12-20. doi: 10.1097/NCC.0000000000000843. PMID 32675630
- [Background] Blackburn L, Hill C, Lindsey AL, Sinnott LT, Thompson K, Quick A. Effect of Foot Reflexology and Aromatherapy on Anxiety and Pain During Brachytherapy for Cervical Cancer. Oncol Nurs Forum. 2021 May 1;48(3):265-276. doi: 10.1188/21.ONF.265-276. PMID 33855996
- [Background] Pascoe MC, Bauer IE. A systematic review of randomised control trials on the effects of yoga on stress measures and mood. J Psychiatr Res. 2015 Sep;68:270-82. doi: 10.1016/j.jpsychires.2015.07.013. Epub 2015 Jul 13. PMID 26228429
- [Background] Schmalzl L, Powers C, Zanesco AP, Yetz N, Groessl EJ, Saron CD. The effect of movement-focused and breath-focused yoga practice on stress parameters and sustained attention: A randomized controlled pilot study. Conscious Cogn. 2018 Oct;65:109-125. doi: 10.1016/j.concog.2018.07.012. Epub 2018 Aug 9. PMID 30099318
- [Background] Danhauer SC, Addington EL, Cohen L, Sohl SJ, Van Puymbroeck M, Albinati NK, Culos-Reed SN. Yoga for symptom management in oncology: A review of the evidence base and future directions for research. Cancer. 2019 Jun 15;125(12):1979-1989. doi: 10.1002/cncr.31979. Epub 2019 Apr 1. PMID 30933317
- [Background] Dhruva A, Miaskowski C, Abrams D, Acree M, Cooper B, Goodman S, Hecht FM. Yoga breathing for cancer chemotherapy-associated symptoms and quality of life: results of a pilot randomized controlled trial. J Altern Complement Med. 2012 May;18(5):473-9. doi: 10.1089/acm.2011.0555. Epub 2012 Apr 23. PMID 22525009
- [Background] Banerjee B, Vadiraj HS, Ram A, Rao R, Jayapal M, Gopinath KS, Ramesh BS, Rao N, Kumar A, Raghuram N, Hegde S, Nagendra HR, Prakash Hande M. Effects of an integrated yoga program in modulating psychological stress and radiation-induced genotoxic stress in breast cancer patients undergoing radiotherapy. Integr Cancer Ther. 2007 Sep;6(3):242-50. doi: 10.1177/1534735407306214. PMID 17761637
- [Background] Akkuzu G, Kurt G, Guvenc G, Kok G, Simsek S, Dogrusoy S, Ayhan A. Learning Needs of Gynecologic Cancer Survivors. J Cancer Educ. 2018 Jun;33(3):544-550. doi: 10.1007/s13187-016-1118-y. PMID 27743314
- [Background] Faravel K, Huteau ME, Jarlier M, de Forges H, Meignant L, Senesse P, Norton J, Jacot W, Stoebner A. Importance of Patient Education for At-home Yoga Practice in Women With Hormonal Therapy-induced Pain During Adjuvant Breast Cancer Treatment: A Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211063791. doi: 10.1177/15347354211063791. PMID 34939444
- [Background] Vieira JS, de Souza GR, Kalil-Cutti B, Giusti-Paiva A, Vilela FC. Post-traumatic stress disorder increases pain sensitivity by reducing descending noradrenergic and serotoninergic modulation. Behav Brain Res. 2021 Aug 6;411:113367. doi: 10.1016/j.bbr.2021.113367. Epub 2021 May 14. PMID 34000338
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Lesage FX, Berjot S, Deschamps F. Psychometric properties of the French versions of the Perceived Stress Scale. Int J Occup Med Environ Health. 2012 Jun;25(2):178-84. doi: 10.2478/S13382-012-0024-8. Epub 2012 Apr 19. PMID 22528542
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Sovik R. The science of breathing--the yogic view. Prog Brain Res. 2000;122:491-505. doi: 10.1016/s0079-6123(08)62159-7. No abstract available. PMID 10737079
- [Derived] Faravel K, Demontoy S, Jarlier M, De-Meric-de-Bellefon M, Cantaloube M, Laboureur E, Meignant L, Del Rio M, Guerdoux E. Impact of an educational physiotherapy-yoga intervention on perceived stress in women treated with brachytherapy for cervical cancer: a randomised controlled mixed study protocol (KYOCOL). BMJ Open. 2025 Jun 4;15(6):e098570. doi: 10.1136/bmjopen-2024-098570. PMID 40467316
- See also: https://www.e-cancer.fr/Patients-et-proches/Les-cancers/Cancer-du-col-de-l-uterus/Quelques-chiffres — https://www.e-cancer.fr/Patients-et-proches/Les-cancers/Cancer-du-col-de-l-uterus/Quelques-chiffres
- See also: https://www.researchgate.net/publication/355647077_Music_Therapy_to_Alleviate_Anxiety_in_Cervical_Brachytherapy_-_Do_We_Change_a_Tune_A_Randomized_Single_Institute_Study — https://www.researchgate.net/publication/355647077_Music_Therapy_to_Alleviate_Anxiety_in_Cervical_Brachytherapy_-_Do_We_Change_a_Tune_A_Randomized_Single_Institute_Study
- See also: https://www.researchgate.net/publication/270634351_Effects_of_music_relaxation_video_on_pain_and_anxiety_for_women_with_gynaecological_cancer_receiving_intracavitary_brachytherapy_a_randomised_controlled_trial — https://www.researchgate.net/publication/270634351_Effects_of_music_relaxation_video_on_pain_and_anxiety_for_women_with_gynaecological_cancer_receiving_intracavitary_brachytherapy_a_randomised_controlled_trial